CLINICAL TRIAL: NCT01153061
Title: Endoscopic Closure of Tracheoesophageal Fistulas With a Cardiac Septal Defect Occluder
Brief Title: Endoscopic Closure of Tracheoesophageal Fistulas With Occluder Device
Acronym: TEFGoreHelex
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated because the rate of prothesis dislocation was too high.
Sponsor: University of Sao Paulo (Other)
Collaborators: InCor Heart Institute (Other); W.L.Gore & Associates (Industry)
Responsible Party: Principal Investigator, Miguel L. Tedde, MD, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USP-0201/10-TEF
Record Dates: First submitted 2010-06-08; First posted 2010-06-29 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Acquired Tracheo-esophageal Fistula
MeSH Terms: interventions — Septal Occluder Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fistula closure with occluder (Experimental): Patients with benign tracheoesophageal fistulas will be submitted to the correction with the occluder.
  Interventions: Device: Fistula closure with Gore Helex Septal Occluder; Device: Gore Helex Septal Occluder

INTERVENTIONS:
Device: Fistula closure with Gore Helex Septal Occluder — The occluder will be released at the tracheoesophageal fistoulous traject through endoscopic procedures
Device: Gore Helex Septal Occluder — Fistula closure with endoscopic release of occluder in the fistula traject.

SUMMARY:
Endoscopic closure of tracheoesophageal fistulas with a device used for closure of cardiac septal defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14 years old
* Benign tracheoesophageal fistulas identified through bronchoscopy;

Exclusion Criteria:

* Malign neoplasia
* Current mechanical ventilation
* Immunosuppressed
* Current local inflammatory process at fistulas borders
* Other clinical risk factors

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Closure of tracheoesophageal fistulas with the Gore Helex Septal Occluder | 6 months
  The closure will be confirmed by endoscopic or bronchoscopic observation of the fistula at regular intervals: one week, two weeks, and four weeks after implant of the occluder.
  A thorax CT scan will ascertain correct positioning and stability of the occluder.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L Tedde, MD, PhD, Principal Investigator — Heart Institute (InCor)-HC of the Sao Paulo University Medica School
Locations (1):
- Heart Institute (InCor)-Clinics Hospital Sao Paulo University Medical School, São Paulo, São Paulo, Brazil